CLINICAL TRIAL: NCT06597877
Title: CT Temporal Bone Anatomical Variations
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nihal Samal Sayed, Nehal Kamal Sayed, Assiut University
Other Study IDs: CT Temporal bone variations
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Temporal Bone Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Radiation: CT — Patients with unilateral ear pathology will be randomly assigned to do CT temporal bone, The presence of five variants was determined. These variants were: a high dehiscent jugular bulb, an anteriorly located sigmoid sinus, a deep sinus tympani, an enlarged cochlear aqueduct, and an enlarged internal auditory meatus (IAM). A GE LightSpeed 16, four-slice, helical CT scanner (Fairfield, Connecticut, USA) was used for all patients. The scan parameters were as follows: 1 mm slices, smart Ma (50-250 Ma), 120 kV, 0.8-second rotation time, 0.562:1 pitch factor, and 5.62 mm rotation speed. All scans covered an area from 1 cm inferior to the mastoid tip to 1 cm superior to the petrous temporal bone.

SUMMARY:
This study aimed to identify the prevalence of normal variations of temporal bone anatomy on high-resolution CT imaging and discuss their clinical importance

DETAILED DESCRIPTION:
The temporal bone has a difficult anatomical structure for otologists and radiologists.In addition to its anatomical complexity, variations in the three-dimensional relationships of structures within the temporal bone need additional attention. The assessment of these relationships is of primary importance in diagnosis, treatment planning, and preoperative management. High-resolution computed tomography (CT) helps locate the anatomical structures within the temporal bone. Preoperative knowledge of the courses of vascular structures within and neighboring the temporal bone is of primary importance. If not detected preoperatively, variations in the localizations of the vascular structures may lead to disastrous consequences during surgery. The surgically important positions of the vascular structures that are generally accepted as normal variants are, High-resolution CT has made it possible for clinicians to study middle- and inner-ear pathology before undertaking surgery. This is particularly useful when the disease has altered the anatomy, resulting in complications such as a lateral canal fistula and facial canal or tegmen erosion there have been several studies reporting the value of high-resolution CT for investigations of cholesteatoma, temporal bone tumors, and congenital anomalies studies on the prevalence of normal anatomical variations of the temporal bone as the use of high-resolution CT imaging for temporal bone investigations is now widespread, it is necessary for the investigating otologist to be aware of common anatomical variations and their clinical implications

ELIGIBILITY:
Inclusion Criteria:

- All adult patients presented with any middle ear pathology indicated for temporal bone radiological evaluation and were willing to participate in the study

Exclusion Criteria:

- 1- patients with temporal bone neoplastic disorders distorting normal temporal bone anatomy.

2- Extensive trauma to the temporal bone 3- Patients with congenital anomalies and craniofacial disproportions 4- Patients with mastoid surgery 5- Patients in whom radiological evaluation is contraindicated

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unilateral ear pathology will be randomly assigned to do CT temporal bone, The presence of five variants was determined. These variants were: a high dehiscent jugular bulb, an anteriorly located sigmoid sinus, a deep sinus tympani, an enlarged cochlear aqueduct, and an enlarged internal auditory meatus (IAM). A GE LightSpeed 16, four-slice, helical CT scanner (Fairfield, Connecticut, USA) was used for all patients. The scan parameters were as follows: 1 mm slices, smart Ma (50-250 Ma), 120 kV, 0.8-second rotation time, 0.562:1 pitch factor, and 5.62 mm rotation speed. All scans covered an area from 1 cm inferior to the mastoid tip to 1 cm superior to the petrous temporal bone.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation of the anatomical variations of the Temporal bone | Baseline
  This study aimed to identify the prevalence of normal variations of temporal bone anatomy on high-resolution CT imaging and discuss their clinical importance This study aimed to identify the prevalence of normal variations of temporal bone anatomy on high-resolution CT imaging and discuss their clinical importance This study aimed to identify the prevalence of normal variations of temporal bone anatomy on high-resolution CT imaging and discuss their clinical importance

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud Roshdy, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walshe P, McConn Walsh R, Brennan P, Walsh M. The role of computerized tomography in the preoperative assessment of chronic suppurative otitis media. Clin Otolaryngol Allied Sci. 2002 Apr;27(2):95-7. doi: 10.1046/j.1365-2273.2002.00538.x. PMID 11994113
- [Background] Visvanathan V, Morrissey MS. Anatomical variations of the temporal bone on high-resolution computed tomography imaging: how common are they? J Laryngol Otol. 2015 Jul;129(7):634-7. doi: 10.1017/S0022215115001115. Epub 2015 Jun 15. PMID 26072959
- [Background] Atilla S, Akpek S, Uslu S, Ilgit ET, Isik S. Computed tomographic evaluation of surgically significant vascular variations related with the temporal bone. Eur J Radiol. 1995 May;20(1):52-6. doi: 10.1016/0720-048x(95)00619-2. PMID 7556255
- [Background] Tatlipinar A, Tuncel A, Ogredik EA, Gokceer T, Uslu C. The role of computed tomography scanning in chronic otitis media. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):33-8. doi: 10.1007/s00405-011-1577-z. Epub 2011 Mar 24. PMID 21431950
- [Background] Jackler RK, Dillon WP, Schindler RA. Computed tomography in suppurative ear disease: a correlation of surgical and radiographic findings. Laryngoscope. 1984 Jun;94(6):746-52. doi: 10.1288/00005537-198406000-00004. PMID 6727511